CLINICAL TRIAL: NCT05802459
Title: Prospective Evaluation of the Functional Status of Jejunoplasty and Coloplasty in Patients Undergoing Complex Esophageal Reconstruction and Its Impact on Quality of Life (CEREC)
Brief Title: Evaluation of the Functional Status of Jejunoplasty and Coloplasty and Its Impact on Quality of Life (CEREC)
Acronym: CEREC
Status: Recruiting | Type: Observational
Sponsor: Hospital Universitari de Bellvitge (Other)
Responsible Party: Principal Investigator, Mònica Miró Martín, Associate surgeon and specialist in Upper Gastrointestinal surgery. PhD, MD., Hospital Universitari de Bellvitge
Other Study IDs: CEREC-2022
Record Dates: First submitted 2023-03-07; First posted 2023-04-06 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-03

CONDITIONS: Quality of Life; Dysphagia
Keywords: Esophageal reconstruction; Quality of life; Coloplasty; Jejunoplasty; Dysphagia
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing complex esophageal reconstruction: All the patients who are candidates for complex esophageal reconstruction performed by the Complex Esophageal Reconstruction Functional Unit of the Bellvitge University Hospital (UREC-HUB), during the study period.
  Interventions: Other: EORTC QLQ-C30; Other: EORTC QLQ-OG25; Other: GIQLI; Other: SWAL QoL; Procedure: Videofluoroscopy

INTERVENTIONS:
Other: EORTC QLQ-C30 — central generic questionnaire associated with different disease specific modules
Other: EORTC QLQ-OG25 — module to assess the quality of life in patients with esophagogastric disease.
Other: GIQLI — Gastrointestinal Quality of Life Index. It is a gastrointestinal quality of life scale.
Other: SWAL QoL — Swallowing Quality of Life questionnaire. This is a quality of life and quality of attention questionnaire for patients with oropharyngeal dysphagia.
Procedure: Videofluoroscopy — It consists of 14 items that represent the oral and pharyngeal function observed in the VDF. It allows to quantify the severity of dysphagia.

SUMMARY:
The goal of this prospective population-based cohort study is to assess:

* The evolution of the functional status of patients undergoing complex esophageal reconstruction
* Its impact on quality of life, depending on the type of conduit performed.

Participants

* Will be asked to complete different quality of life questionnaires during every follow-up visit
* Will undergo additional tests to assess functionality

DETAILED DESCRIPTION:
-General Justification: In recent years, esophageal reconstruction has been a great surgical challenge for the multidisciplinary teams in charge of carrying out this complex technique, associated with high morbidity and a high impact on the quality of life and functional status of patients.

One of the most important aspects of this surgery is the type of conduit used to restore digestive transit. Classically, gastroplasty has been the technique of choice due to its lower morbidity and mortality and less surgical complexity. On the other hand, in those patients in whom the stomach is not available, a coloplasty or a jejunoplasty is chosen, both of which can be associated with supercharged techniques to improve and ensure good vascular flow.

Currently, there is controversy about which type of conduit to use in the absence of a viable stomach. Since the introduction of microvascular or supercharged techniques, the postoperative results of jejunal grafts are comparable to coloplasty and even gastroplasty according to some authors.

The present study is an initiative of the Complex Esophageal Reconstruction Unit (UREC) of Bellvitge University Hospital (HUB), which aims to compare the different types of conduit used in complex esophageal reconstruction, assessing, in the short and long term, the postoperative functional status and its impact on quality of life through validated test-type tools, as well as carrying out complementary tests that allow evaluating aspects such as swallowing and dysphagia, among others.

* Hypothesis Considering the results of quality of life and functionality in the short and long term, jejunoplasty (free, pedunculated ± supercharged) could be the second technique of choice to perform in the absence of gastric conduit in complex esophageal reconstruction.
* Primary objective:

  1. To determine the differences in the quality of life of patients undergoing complex esophageal reconstruction by jejunoplasty (free, pedunculated ± supercharged) or coloplasty (± supercharged).
  2. To describe the functional evolution of complex esophageal reconstruction by jejunoplasty (free, pedunculated ± supercharged) or coloplasty (± supercharged).
* Study design CEREC-2022 is a prospective population-based cohort study that aims to assess the evolution of the functional status of patients undergoing complex esophageal reconstruction and its impact on quality of life, depending on the type of conduit performed.
* Study population The target population of this study is made up of patients who are candidates for complex esophageal reconstruction performed by the Complex Esophageal Reconstruction Functional Unit of the Bellvitge University Hospital (UREC-HUB), during the study period. All patients who are candidates for complete replacement of the esophagus through reconstruction are presented to the Committee of the Complex Esophageal Reconstruction Functional Unit of the Bellvitge University Hospital (UREC-HUB). After the multidisciplinary assessment, the most appropriate type of surgery for each patient is proposed and the patient receives the information during a scheduled appointment, at this moment the patient is asked to participate in the CEREC-2022 study.
* Main Outcome

  1. Quality of life related to the swallowing function based on the conduit: it will be assessed using the European Organisation for Research and Treatment of Cancer Quality-of-life Questionnaire Core 30 (EORTC QLQ C30), European Organisation for Research and Treatment of Cancer Quality-of-life Questionnaire Oesophago Gastric module 25 (EORTC QLQ OG25), Gastrointestinal quality of life index (GIQLI) and Swallowing quality of life questionnaire (SWAL QoL)
  2. Number (percentage) of patients who present tolerance to the oral intake and need (volume in milliliters) of enteral nutrition depending on the type of conduit.
* Secondary outcome Incidence of dysphagia evaluated by Videofluoroscopy (VDF), Incidence of stenosis of the conduit in the Upper Digestive Endoscopy (UDE), Number (percentage) of dilatations of the conduit, Number (percentage) of patients with esophagitis according to the Los Angeles classification, Nutritional status, Number (percentage) of specific complications of the surgery during admission according to the Esophageal Complication Consensus Group, Number of hospitalizations.
* As this is an observational study of a low-prevalent surgical indication, it is expected to include all patients scheduled for surgery from September 2022 to September 2025.
* The follow-up of each patient included in the study will end 3 years after the intervention when the End of Study visit will be carried out.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 18 years of age) and of both gender.
* Candidates for complete esophageal reconstruction with cervical anastomosis, regardless of the etiology of the esophagectomy.
* Decision to indicate a coloplasty (+/- supercharged) or jejunoplasty (free, pedunculated +/- supercharged) as surgical technique after evaluation by the UREC Committee.
* Acceptance to participate in the study and comply with the program of procedures (schedule of visits).
* Signing of the informed consent.

Exclusion Criteria:

* Patients who withdraw their informed consent at any time during the course of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population of this study is made up of patients who are candidates for complex esophageal reconstruction performed by the Complex Esophageal Reconstruction Functional Unit of the Bellvitge University Hospital (UREC-HUB), during the study period.
  All patients who are candidates for complete replacement of the esophagus through reconstruction are presented to the Committee of the Complex Esophageal Reconstruction Functional Unit of the Bellvitge University Hospital (UREC-HUB). After the multidisciplinary assessment, the most appropriate type of surgery for each patient is proposed and the patient receives the information during a scheduled appointment, at this moment the patient is asked to participate in the CEREC-2022 study.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2022-12-15 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Quality of life related to the swallowing function assessed using the EORTC QLQ OG25, EORTC QLQ C30, GIQLI and SWAL QoL questionnaire. | The follow-up of each patient included in the study will end 3 years after the intervention when the End of Study visit will be carried out.
  This study aims to determine the differences in the quality of life of patients undergoing complex esophageal reconstruction by jejunoplasty (free, pedunculated ± supercharged) or coloplasty (± supercharged) using the following questionnaires:
  * European Organisation for Research and Treatment of Cancer Quality-of-life Questionnaire Core 30 (EORTC QLQ C30): All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
  * European Organisation for Research and Treatment of Cancer Quality-of-life Questionnaire Oesophago Gastric module 25 (EORTC QLQ OG25): All of the scales and single-item measures range in score from 0 to 100. A high score for all the scales and single-items represents a high level of symptomatology or problems.
  * Gastrointestinal quality of life index (GIQLI): scale range from 0-144
  * Swallowing quality of life questionnaire (SWAL QoL): scale range from 0-100
Number (percentage) of patients who present tolerance to the oral intake and need (volume in milliliters) of enteral nutrition depending on the type of conduit. | The follow-up of each patient included in the study will end 3 years after the intervention when the End of Study visit will be carried out.
  This study aims to describe the functional evolution of complex esophageal reconstruction by jejunoplasty (free, pedunculated ± supercharged) or coloplasty (± supercharged).

SECONDARY OUTCOMES:
Incidence of dysphagia | The follow-up of each patient included in the study will end 3 years after the intervention when the End of Study visit will be carried out.
  Incidence of dysphagia evaluated by Videofluoroscopic (VDF) using the following scales:
  * Videofluoroscopic dysphagia scale (VDS)
  * Dysphagia outcome and severity scale(DOSS)
  * Penetration-aspiration scale(PAS)
Incidence of stenosis of the conduit | The follow-up of each patient included in the study will end 3 years after the intervention when the End of Study visit will be carried out.
  Incidence of stenosis of the conduit in the Upper Digestive Endoscopy (UDE) that requires some therapeutic maneuver (dilatation), which is carried out during the follow-up visits: one year, two and three years.
Number (percentage) of dilatations of the conduit | The follow-up of each patient included in the study will end 3 years after the intervention when the End of Study visit will be carried out.
  Number (percentage) of dilatations of the conduit, per patient, carried out during the UDE within the follow-up visits: one year, two and three years.
Number (percentage) of patients with esophagitis | The follow-up of each patient included in the study will end 3 years after the intervention when the End of Study visit will be carried out.
  Number (percentage) of patients with esophagitis according to the Los Angeles classification evidenced in any of the UDE performed during the follow-up visits: one year, two and three years.
Number (percentage) of patients with chronic diarrhea | The follow-up of each patient included in the study will end 3 years after the intervention when the End of Study visit will be carried out.
  Number (percentage) of patients with chronic diarrhea during follow-up
Body Mass Index | The follow-up of each patient included in the study will end 3 years after the intervention when the End of Study visit will be carried out.
  Weight and height will be combined to report Body Mass Index (BMI kg/m2) as a measure for indicating nutritional status
Muscle strength measured by Handgrip strength (HGS) dynamometer | The follow-up of each patient included in the study will end 3 years after the intervention when the End of Study visit will be carried out.
  Handgrip strength expressed in Kg and assessed using the reference values for age and sex
Serum albumin value | The follow-up of each patient included in the study will end 3 years after the intervention when the End of Study visit will be carried out.
  Measure of albumin/prealbumin in blood tests for assessment of nutritional status. Normal value: 34 - 54 g/L
Mean 'time of need for enteral nutrition and oral nutrition supplements' | The follow-up of each patient included in the study will end 3 years after the intervention when the End of Study visit will be carried out.
  Mean 'time of need for enteral nutrition and oral nutrition supplements' during the post-surgical follow-up period.
Volume of enteral nutrition required | The follow-up of each patient included in the study will end 3 years after the intervention when the End of Study visit will be carried out.
  Volume of enteral nutrition required during the post-surgical follow-up period.
Number of hospitalizations | The follow-up of each patient included in the study will end 3 years after the intervention when the End of Study visit will be carried out.
  Number of hospitalizations, for any reason, during the post-surgical follow-up period.
Number (percentage) of specific complications of the surgery during admission according to the Esophageal Complication Consensus Group (ECCG) | The follow-up of each patient included in the study will end 3 years after the intervention when the End of Study visit will be carried out.
  Number (percentage) of specific complications of the surgery during admission according to the Esophageal Complication Consensus Group (ECCG) (20), highlighting anastomotic dehiscence, surgical site infection, bleeding, need for reintervention, ischaemia of the graft (up to 90 ±3 days after surgery). Number (percentage) of complications according to the Clavien-Dindo classification (21) and Comprehensive Complication Index.
Mortality | The follow-up of each patient included in the study will end 3 years after the intervention when the End of Study visit will be carried out.
  Number (percentage) of deaths related to esophageal reconstruction (Up to 90 ±3 days after surgery).

CONTACTS AND LOCATIONS:
Overall Officials: Leandre Farran, Study Director — Bellvitge University Hospital
Locations (1):
- Hospital Uversitari de Bellvitge, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bothereau H, Munoz-Bongrand N, Lambert B, Montemagno S, Cattan P, Sarfati E. Esophageal reconstruction after caustic injury: is there still a place for right coloplasty? Am J Surg. 2007 Jun;193(6):660-4. doi: 10.1016/j.amjsurg.2006.08.074. PMID 17512272
- [Background] Farran-Teixido L, Miro-Martin M, Biondo S, Conde-Mourino R, Bettonica-Larranaga C, Aranda Danso H, Sans-Segarra M, Rafecas-Renau A. [Second time esophageal reconstruction surgery: coloplasty and gastroplasty]. Cir Esp. 2008 May;83(5):242-6. doi: 10.1016/s0009-739x(08)70561-x. Spanish. PMID 18448026
- [Background] Irino T, Tsekrekos A, Coppola A, Scandavini CM, Shetye A, Lundell L, Rouvelas I. Long-term functional outcomes after replacement of the esophagus with gastric, colonic, or jejunal conduits: a systematic literature review. Dis Esophagus. 2017 Dec 1;30(12):1-11. doi: 10.1093/dote/dox083. PMID 28881882
- [Background] Jacobs M, Macefield RC, Elbers RG, Sitnikova K, Korfage IJ, Smets EM, Henselmans I, van Berge Henegouwen MI, de Haes JC, Blazeby JM, Sprangers MA. Meta-analysis shows clinically relevant and long-lasting deterioration in health-related quality of life after esophageal cancer surgery. Qual Life Res. 2014 May;23(4):1097-115. doi: 10.1007/s11136-013-0545-z. Epub 2013 Oct 16. PMID 24129668
- [Background] Miro M, Farran L, Estremiana F, Miquel J, Escalante E, Aranda H, Bettonica C, Galan M. Does gastric conditioning decrease the incidence of cervical oesophagogastric anastomotic leakage? Cir Esp (Engl Ed). 2018 Feb;96(2):102-108. doi: 10.1016/j.ciresp.2017.11.012. Epub 2018 Feb 17. English, Spanish. PMID 29459004
- [Background] Lamas S, Azuara D, de Oca J, Sans M, Farran L, Alba E, Escalante E, Rafecas A. Time course of necrosis/apoptosis and neovascularization during experimental gastric conditioning. Dis Esophagus. 2008;21(4):370-6. doi: 10.1111/j.1442-2050.2007.00772.x. PMID 18477261
- [Background] Farran Teixidor L, Vinals Vinals JM, Miro Martin M, Higueras Sune C, Bettonica Larranaga C, Aranda Danso H, Lopez Ojeda A, Rafecas Renau A. [Supercharged ileocoloplasty: an option for complex oesophageal reconstructions]. Cir Esp. 2011 Feb;89(2):87-93. doi: 10.1016/j.ciresp.2010.10.009. Epub 2011 Feb 1. Spanish. PMID 21277572
- [Background] Ochsner A, Owens N. Anterothoracic Oesophagoplasty for Impermeable Stricture of the Oesophagus. Ann Surg. 1934 Dec;100(6):1055-91. doi: 10.1097/00000658-193412000-00002. No abstract available. PMID 17856421
- [Background] Jiang S, Guo C, Zou B, Xie J, Xiong Z, Kuang Y, Tang J. Comparison of outcomes of pedicled jejunal and colonic conduit for esophageal reconstruction. BMC Surg. 2020 Jul 16;20(1):156. doi: 10.1186/s12893-020-00810-y. PMID 32677925
- [Background] Luan A, Hunter CL, Crowe CS, Lee GK. Comparison of Outcomes of Total Esophageal Reconstruction With Supercharged Jejunal Flap, Colonic Interposition, and Gastric Pull-up. Ann Plast Surg. 2018 May;80(5S Suppl 5):S274-S278. doi: 10.1097/SAP.0000000000001471. PMID 29634501
- [Background] Blackmon SH, Correa AM, Skoracki R, Chevray PM, Kim MP, Mehran RJ, Rice DC, Roth JA, Swisher SG, Vaporciyan AA, Yu P, Walsh GL, Hofstetter WL. Supercharged pedicled jejunal interposition for esophageal replacement: a 10-year experience. Ann Thorac Surg. 2012 Oct;94(4):1104-11; discussion 1111-3. doi: 10.1016/j.athoracsur.2012.05.123. Epub 2012 Aug 29. PMID 22939245
- [Background] Yasuda T, Shiozaki H. Esophageal reconstruction using a pedicled jejunum with microvascular augmentation. Ann Thorac Cardiovasc Surg. 2011;17(2):103-9. doi: 10.5761/atcs.ra.10.01648. PMID 21597405
- [Background] Yang YS, Shang QX, Yuan Y, Wu XY, Hu WP, Chen LQ. Comparison of Long-term Quality of Life in Patients with Esophageal Cancer after Ivor-Lewis, Mckeown, or Sweet Esophagectomy. J Gastrointest Surg. 2019 Feb;23(2):225-231. doi: 10.1007/s11605-018-3999-z. Epub 2018 Oct 8. PMID 30298418
- [Background] Stephens EH, Gaur P, Hotze KO, Correa AM, Kim MP, Blackmon SH. Super-Charged Pedicled Jejunal Interposition Performance Compares Favorably With a Gastric Conduit After Esophagectomy. Ann Thorac Surg. 2015 Aug;100(2):407-13. doi: 10.1016/j.athoracsur.2015.03.040. Epub 2015 Jun 20. PMID 26101096
- [Background] Mahajan NN, Lee MK, Yost KJ, Pierson KE, Viehman JK, Allen MS, Cassivi SD, Nichols FC, Reisenauer JS, Shen KR, Wigle DA, Blackmon SH. Preliminary Normative Standards of the Mayo Clinic Esophagectomy CONDUIT Tool. Mayo Clin Proc Innov Qual Outcomes. 2019 Nov 22;3(4):429-437. doi: 10.1016/j.mayocpiqo.2019.07.008. eCollection 2019 Dec. PMID 31993561
- [Background] Lee MK, Yost KJ, Pierson KE, Schrandt AJ, Skaare BJ, Blackmon SH. Standard setting for a novel esophageal conduit questionnaire: CONDUIT Report Card. J Patient Rep Outcomes. 2018 Oct 24;2(1):51. doi: 10.1186/s41687-018-0073-2. PMID 30467674
- [Background] Lagergren P, Fayers P, Conroy T, Stein HJ, Sezer O, Hardwick R, Hammerlid E, Bottomley A, Van Cutsem E, Blazeby JM; European Organisation for Research Treatment of Cancer Gastrointestinal and Quality of Life Groups. Clinical and psychometric validation of a questionnaire module, the EORTC QLQ-OG25, to assess health-related quality of life in patients with cancer of the oesophagus, the oesophago-gastric junction and the stomach. Eur J Cancer. 2007 Sep;43(14):2066-73. doi: 10.1016/j.ejca.2007.07.005. Epub 2007 Aug 15. PMID 17702567
- [Background] Low DE, Alderson D, Cecconello I, Chang AC, Darling GE, D'Journo XB, Griffin SM, Holscher AH, Hofstetter WL, Jobe BA, Kitagawa Y, Kucharczuk JC, Law SY, Lerut TE, Maynard N, Pera M, Peters JH, Pramesh CS, Reynolds JV, Smithers BM, van Lanschot JJ. International Consensus on Standardization of Data Collection for Complications Associated With Esophagectomy: Esophagectomy Complications Consensus Group (ECCG). Ann Surg. 2015 Aug;262(2):286-94. doi: 10.1097/SLA.0000000000001098. PMID 25607756
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Background] Kim J, Oh BM, Kim JY, Lee GJ, Lee SA, Han TR. Validation of the videofluoroscopic dysphagia scale in various etiologies. Dysphagia. 2014 Aug;29(4):438-43. doi: 10.1007/s00455-014-9524-y. PMID 24658847
- [Background] O'Neil KH, Purdy M, Falk J, Gallo L. The Dysphagia Outcome and Severity Scale. Dysphagia. 1999 Summer;14(3):139-45. doi: 10.1007/PL00009595. PMID 10341109
- [Background] Rosenbek JC, Robbins JA, Roecker EB, Coyle JL, Wood JL. A penetration-aspiration scale. Dysphagia. 1996 Spring;11(2):93-8. doi: 10.1007/BF00417897. PMID 8721066
- [Background] Clave P, Arreola V, Velasco M, Quer M, Castellvi JM, Almirall J, Garcia Peris P, Carrau R. [Diagnosis and treatment of functional oropharyngeal dysphagia. Features of interest to the digestive surgeon]. Cir Esp. 2007 Aug;82(2):62-76. doi: 10.1016/s0009-739x(07)71672-x. Spanish. PMID 17785140
- [Background] Crary MA, Mann GD, Groher ME. Initial psychometric assessment of a functional oral intake scale for dysphagia in stroke patients. Arch Phys Med Rehabil. 2005 Aug;86(8):1516-20. doi: 10.1016/j.apmr.2004.11.049. PMID 16084801
- [Background] Schiller LR, Pardi DS, Sellin JH. Chronic Diarrhea: Diagnosis and Management. Clin Gastroenterol Hepatol. 2017 Feb;15(2):182-193.e3. doi: 10.1016/j.cgh.2016.07.028. Epub 2016 Aug 2. PMID 27496381
- [Background] Konradsson M, van Berge Henegouwen MI, Bruns C, Chaudry MA, Cheong E, Cuesta MA, Darling GE, Gisbertz SS, Griffin SM, Gutschow CA, van Hillegersberg R, Hofstetter W, Holscher AH, Kitagawa Y, van Lanschot JJB, Lindblad M, Ferri LE, Low DE, Luyer MDP, Ndegwa N, Mercer S, Moorthy K, Morse CR, Nafteux P, Nieuwehuijzen GAP, Pattyn P, Rosman C, Ruurda JP, Rasanen J, Schneider PM, Schroder W, Sgromo B, Van Veer H, Wijnhoven BPL, Nilsson M. Diagnostic criteria and symptom grading for delayed gastric conduit emptying after esophagectomy for cancer: international expert consensus based on a modified Delphi process. Dis Esophagus. 2020 Apr 15;33(4):doz074. doi: 10.1093/dote/doz074. PMID 31608938